CLINICAL TRIAL: NCT04760366
Title: Effects of Fascial-muscular Lengthening Therapy on Tight Iliopsoas Muscle in the Patients With Chronic Low Back Pain.
Brief Title: Fascial-muscular Lengthening Therapy in the Patients With Chronic Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00766 Najia Zainab
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Chronic Low Back Pain
Keywords: FMLT; Chronic LWP; ROM; ODI; NPRS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental) (Experimental): Patients in this group will receive interventional therapy through fascial- muscular lengthening therapy .Patients in this group will also receive the conventional therapy
  Interventions: Other: fascial- muscular lengthening therapy; Other: the conventional therapy
- Group B: Conventional treatment (Other): Patients in this group will receive the conventional therapy
  Interventions: Other: Stretching's of iliopsoas muscle; Other: the conventional therapy

INTERVENTIONS:
Other: fascial- muscular lengthening therapy — Patients in this group will receive interventional therapy
  To perform this technique:
  1. Have the patient in side lying position
  2. Hip is maximally flexed to shorten the iliopsoas muscle.
  3. Therapist fingers should be on to the targeted area.
  4. Apply gentle pressure in upward direction.
  5. While maintain the pressure, stretch the muscle by moving the hip in extension through full ROM.
  6. Therapist will maintain the pressure in opposing direction. This is considered as one pass. This technique is performed bilaterally. Patients in this group will also receive the conventional therapy which will include:
     * Hot pack for 15 minutes.
     * Myofascial release of iliopsoas.
     * TENS for 15 minutes.
  Arms: Group A (Experimental)
Other: Stretching's of iliopsoas muscle — Patients in this group will receive the interventional therapy which will include:
  Stretching's of iliopsoas muscle which can be done in two positions:
  1. modified lunge position.
  2. The prone stretch.
  Patients in this group will also receive the conventional therapy which will include:
  * Hot pack for 15 minutes.
  * Myofascial release of iliopsoas
  * TENS for 15 minutes.
  Arms: Group B: Conventional treatment
Other: the conventional therapy — the conventional therapy

SUMMARY:
The purpose of this study is to assess and evaluate tight iliopsoas muscle in patients with chronic low back pain and to increase hip flexor flexibility in the patients with chronic low back pain by using the technique of manual fascial-muscular lengthening therapy .

DETAILED DESCRIPTION:
Chronic low back pain is one of the the most prevalent complaint in the patients. Low back pain is affecting the population socially and economically, and it is also a leading public health problem, being the very common reason for absentees from work . Living with chronic low back pain leads to not only physiological but also psychological modifications. Low back pain is associated with many biomechanical factors that must not be ignored because in some cases mechanical loading results in acute disc prolapse and can also cause low back pain

The iliopsoas muscle is the primary and the most strongest hip flexor and it plays vital role in the stability of the lumbar spine for axial compression but it has very little movement function on the lumbar spine. Like other postural muscles it functions as stabilizer, and for spinal stability iliopsoas activity is essential although iliopsoas can only produce minimum movements in the sagittal plane. It is assumed that muscle weakness and other structural factors can cause low back pain and activity limitation. As the psoas muscle is the postural muscles so it also has tendency to become tight Psoas muscle tightness is responsible for causing back pain by inhibiting the lumbar and SI-joint range of motion but in the literature there is more focus on hamstring tightness rather than on iliopsoas tightness .The psoas muscle should not be ignored when evaluating and treating low back pain. because iliopsoas muscle tightness can also manifest low back pain, giving the symptoms of lumbosacral region pain, contralateral gluteal region pain and radiating pain in contralateral leg.

There has been a lot of procedures which are used to increase muscle flexibility of tight hip flexors e.g. Active and passive stretching , manual fascial-muscular lengthening therapy , a form of Active Release Technique, proprioceptive neuromuscular facilitation soft tissue mobilization and strengthening of psoas muscle.

Stretching programmers are often part of Physical Therapy treatment plan to increase muscle flexibility. A study done on Passive versus active stretching of hip flexor muscles in subjects with limited hip extension. concluded that active and passive stretching of tight hip flexors will increase the flexibility of hip flexors and range of motion in patient with low back pain

A study on "Low Back Pain with Psoas Tightness" in 2012 and concluded that the low back pain begins when there's irritation in the psoas muscle and he used soft tissue mobilization techniques and strengthening program of hip flexors to treat chronic low back pain which resulted in diminished back pain.

A study on The clinical and biomechanical effects of fascial- muscular lengthening therapy on tight hip flexor patients with and without low back pain in 2014 and concluded that by using fascial-muscular lengthening therapy there was a reduction in low back pain. There was increase in the range of passive hip extension and there was also significant decrease in iliopsoas tightness in the patients with or without low back pain.

A study on Immediate effect of application of the pressure technique to the psoas major on lumbar lordosis in 2018 in which mechanical pressure, which is similar to fascial-muscular lengthening therapy, was applied to the psoas major muscle and concluded that pressure technique reduced psoas major stiffness along with reducing lumbar extension on every segment.

ELIGIBILITY:
Inclusion Criteria:

* • The study includes female patients with chronic low back pain.

  * The study includes patients from the age group of 25 years and 45.
  * The study includes patients with low back pain for more than 3 months.
  * The study includes patients with chronic bilateral tight hip flexors which will assessed through Thomas Test
  * Pain in flexion bias

Exclusion Criteria:

* • The study excludes male patients.

  * No history of serious underlying pathology, nerve root compromise, structural deformities, genetic spinal disorders or previous spinal surgery

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — • The study includes female patients with chronic low back pain
Enrollment: 76 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6th day
  This scale will be used for assessing low back pain before and after treatment.0 no pain 1-4 mild pain 5-7 moderate and 8-10 sever pain. Baseline,6th day
For disability: Oswestry Disability Index (ODI) | 6th day
  Tool used to assess disability related to pain in individuals with acute, sub-acute, or chronic LBP. The total score of ODI range from 0 (no disability) to 100 (maximum disability). The ODI score is recommended as a back pain-specific measure of disability. Reliability with ICC= 0.85 and validity=0.77 Baseline,6th day
For tight iliopsoas: Thomas Test. | 6th day
  This test is used to test the flexibility of hip flexors.Baseline,6th day

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Shahid, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No